CLINICAL TRIAL: NCT06255782
Title: A Phase 1/2/3 First-in-Human, Open-Label, Dose-Escalation Study to Evaluate the Safety and Efficacy of a Single Intravenous (IV) Administration of ECUR-506 in Males Less Than 9 Months of Age With Genetically Confirmed Neonatal Onset Ornithine Transcarbamylase (OTC) Deficiency
Brief Title: An Open-label Study to Investigate ECUR-506 in Male Babies Less Than 9 Months of Age With Neonatal Onset OTC Deficiency
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: iECURE, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ECUR-506-OTC-101; OTC HOPE (Other: iECURE, Inc.)
Record Dates: First submitted 2023-12-19; First posted 2024-02-13 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Ornithine Transcarbamylase Deficiency; Ornithine Transcarbamylase Deficiency Disease; Ornithine Carbamoyltransferase Deficiency (Disorder); Urea Cycle Disorders, Inborn
Keywords: Amino Acid Metabolism, Inborn Errors; Ammonia; Brain Diseases; Brain Diseases, Metabolic; Brain Diseases, Metabolic, Inborn; Central Nervous System Diseases; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; High Ammonia; Hyperammonemia; Inborn; Inborn Errors; Liver Disease; Liver Transplant; Metabolism; Metabolic Diseases; Metabolism, Inborn Errors; Neonatal; Nervous System Diseases; NH4; Ornithine; Ornithine Transcarbamylase Deficiency; OTC; OTC Deficiency; OTCD; Transcarbamylase; UCD; Urea Cycle Disorders; X-Linked
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease; Urea Cycle Disorders, Inborn; Amino Acid Metabolism, Inborn Errors; Brain Diseases; Brain Diseases, Metabolic; Brain Diseases, Metabolic, Inborn; Central Nervous System Diseases; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; Hyperammonemia; Liver Diseases; Metabolic Diseases; Metabolism, Inborn Errors; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Dose escalation with dose staggering. Dose selection will be based on an assessment of the totality of the safety and efficacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose Level (Experimental): Participants will receive the Low Dose of ECUR-506 delivered one time via IV Infusion.
  Interventions: Genetic: ECUR-506
- High Dose Level (Experimental): Participants will receive a higher dose of ECUR-506 delivered one time via IV infusion.
  Interventions: Genetic: ECUR-506
- Intermediate Dose Level (Experimental): Additional Cohorts based on recommendations of DMC review of safety and efficacy data.
  Interventions: Genetic: ECUR-506

INTERVENTIONS:
Genetic: ECUR-506 — ECUR-506 is a gene editing treatment delivering a gene encoding the editing enzyme and an OTC gene.

SUMMARY:
Ornithine Transcarbamylase (OTC) deficiency, the most common urea cycle disorder, is an inherited metabolic disorder caused by a genetic defect in a liver enzyme responsible for detoxification of ammonia. Individuals with OTC deficiency can build-up excess levels of ammonia in their blood, potentially resulting in devastating consequences, including cumulative and irreversible neurological damage, coma and death. The severe form of the condition emerges shortly after birth and is more common in boys than girls.

This is a Phase 1/2/3, open-label, multicenter, safety, efficacy, and dose finding study of ECUR-506 in male babies with neonatal onset OTC deficiency. The primary objective of this study is to evaluate the safety, tolerability, and efficacy of up to three dose levels of ECUR-506 following intravenous (IV) administration of a single dose.

DETAILED DESCRIPTION:
The study drug, ECUR-506, is an investigational gene editing therapy. Gene editing is a way to repair, replace, or introduce new copies of genes that don't work. The study drug contains a working copy of the OTC gene that will be delivered by an IV infusion. It also contains a gene to encode the editing enzyme which is the part of the study drug that can cut DNA so that the OTC gene can be inserted. The study drug was designed to introduce a working copy of the OTC gene and a gene to encode the editing enzyme. A gene cannot enter cells by itself, it needs a delivery mechanism to move the gene into the cells. In this study, a commonly used virus called adeno-associated virus (AAV) is used to enter the cells and deliver the genes.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male sex
2. Gestational or adjusted (corrected) gestational age ≥ 37 weeks
3. Age at screening is 24 hours to 7 months
4. Weight ≥ 3.5 kg and ≤ 13.5 kg at screening
5. Has received age-appropriate vaccinations
6. Genetically confirmed OTCD
7. Severe neonatal OTCD defined by hyperammonemic crisis with elevated ammonia level of >560 μmol/L and clinical symptoms within first week of life
8. Current or historical biochemical profile consistent with OTCD
9. Participant's parent(s)/LAR must be able to comprehend and be willing to provide a signed IRB/IEC-approved ICF.

Key Exclusion Criteria:

1. Neonatal diagnosis of severe to profound Hypoxic Ischemic Encephalopathy due to birth injury
2. Requiring urgent liver transplant due to liver failure as assessed by the PI.
3. Contiguous gene deletion involving the OTC gene and including at least the CYBB gene on the telomeric side or the TSPAN7 gene on the centromeric side.
4. Known or suspected major organ injury/dysfunction/anomalies.
5. Vital sign abnormalities
6. Laboratory abnormalities outside of laboratory normal ranges for urinalysis, complete blood count, and comprehensive metabolic panel that are attributable to comorbidities unrelated to OTCD
7. Treatment with any other gene therapy or gene editing therapy
8. Co-enrollment in any other clinical study unless approved by the sponsor.
9. Any condition, that in the opinion of the Investigator, would compromise the safety of the participant or study data
10. Documented vertical transmission of HepA/HepB/HepC
11. Documented in-utero teratogen, substance, and/or alcohol exposure, which in the opinion of the Investigator may increase the participant's risk of developmental delays, congenital anomalies, and/or significant medical complications

Ages: 24 Hours to 7 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Males present with the highest unmet medical need, and in order to reduce the variability of the study population, participants are restricted to the male sex . OTC is primarily inherited in an X-linked recessive pattern, meaning that it mostly affects males, who only have one copy of the X chromosome. Females, who have two X chromosomes, can be carriers of the condition. Some females may experience milder OTC symptoms, or they may have no symptoms.
Enrollment: 8 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (incidence, severity, seriousness, and relatedness) | Over 24 weeks post infusion
  Toxicity is graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Adverse events (AEs) are reported based on clinical laboratory tests, vital signs, physical examinations, Pediatric Neurologist exam parameters, electrocardiograms, and any other medically indicated assessments from the time informed consent is signed through the end of the safety follow-up period.
  AEs are considered to be treatment emergent (TEAE) if they occur or worsen in severity following the administration of the study treatment. TEAEs are considered treatment-related if relationship to study drug is possibly related, probably related, or definitely related.
Urinalysis evaluations | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Toxicity is graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Adverse events (AEs) are reported based on clinical laboratory tests, vital signs, physical examinations, electrocardiograms, and any other medically indicated assessments from the time informed consent is signed through the end of the safety follow-up period.
  AEs are considered to be treatment emergent (TEAE) if they occur or worsen in severity following the administration of the study treatment. TEAEs are considered treatment-related if relationship to study drug is possibly related, probably related, or definitely related.
Achieving normal fasting plasma ammonia levels by EOS | Over 24 weeks post infusion
  Fasting plasma ammonia levels that fall within normal limits for at least 75% of post-dose assessments.
Complete clinical response | Over 24 weeks post infusion
  Discontinuation of scavenger medication for a minimum duration of 28 days without reductions in prescribed daily protein intake during this time period.

SECONDARY OUTCOMES:
Percent liver transduction | Assessed at Week 24
  Pharmacokinetics
Number of hyperammonemic crises (HAC) | Over 24 weeks post infusion
  Pharmacodynamics and Efficacy
qPCR measurement to evaluate the clearance of both vectors in body fluids over time | Over 24 weeks post infusion
  Pharmacokinetics
Scavenger drug dose per body surface area (BSA) | Over 24 weeks post infusion
  Efficacy
Protein allowance g/kg/day | Over 24 weeks post infusion
  Efficacy
Blood urea nitrogen measurements | Over 24 weeks post infusion
  Pharmacodynamics
Fasting plasma ammonia | Over 24 weeks post infusion
  Efficacy

OTHER OUTCOMES:
Serum Neurofilament Light Chain evaluation | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Safety
Number of participants with antibodies to hOTC in blood | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Pharmacodynamics
Number of participants with antibodies to M2PCSK9 in blood | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Pharmacodynamics
Number of participants with antibodies to AAVrh79 in blood | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Pharmacodynamics
Daily ammonia levels during hospitalization requiring ICU care for HAC event | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Pharmacodynamics and Safety
Time to liver transplant from dosing to end of study (EOS) | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Efficacy
Transplant free survival | Time to liver transplant or any-cause death from dosing to EOS
  Efficacy
Overall survival | Time to any-cause death from dosing to EOS
  Efficacy
Number of instances the participant is eligible for medical management adjustments based on iECURE guidance (protein diet or scavenger medication) | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Efficacy
Fasting plasma ammonia, fasting plasma citrulline and fasting plasma glutamine levels | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Pharmacodynamics
Serum PCSK9 | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Pharmacodynamics
Change from baseline at Week 24 post infusion in Bayley Scales of Infant and Toddler Development 4th Ed (BSID-4) for the Cognitive, Language, and Motor scales | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Total Raw Scores, Growth Score Values (GSVs), and Age Equivalent Scores will be analyzed; Raw Scores range 0-162; GSVs range 428-599; Age Equivalent Scores range 1-42 months; a higher score reflects a higher level of skill.
Quality of Life, as measured by the Pediatric QOL inventory Infant Scale (PedsQL-IS) | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Quality of Life
Urinary excretion of phenylacetate metabolites | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Urinary phenylacetate (mcg/mL), urinary phenylacetylglutamine (mcg/mL), urinary phenylacetate/ phenylglutamine ratio.
Urinary excretion of orotic acid metabolites. | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Urinary orotic acid (mmol/ mol creatinine), urinary uracil (mmol/mol creatinine).
Urinary nitrogen to urinary creatinine ratio. | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Urinary nitrogen to urinary creatinine ratio (mg/dL)
Change from baseline at Week 24 post infusion in length. | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Length measured in centimeters.
Change from baseline at Week 24 post infusion in weight. | Assessed as change from baseline at pre-specified timepoints through Week 24 post infusion.
  Weight measured in kilograms.
Assess the potential on target editing by amplicon-seq in liver tissue samples of participants who received ECUR-506. | The following will be assessed at week 24 if liver biopsy tissue sample is sufficient.
  Pharmacodynamics
Assess potential off-target editing with AAV vector ITR insertion by ITR-seq in liver tissue samples of participants who recieved ECUR-506 | The following will be assessed at Week 24 if liver biopsy tissue sample is sufficient.
  Pharmacodynamics
Assess for potential genetic changes in the liver tissue, collected by liver biopsy, through long read sequencing, in participants who have received ECUR-506 | The following will be assessed at Week 24 if liver biopsy tissue sample is sufficient.
  Pharmacodynamics
With an observed genetic safety signal, genetic analysis of Whole Blood DNA may be performed on samples collected and stored at screening and week 24, in the event of an observed genomic safety signal. | Assessed as any difference between screening and week 24 genetic markers, if a genetic safety signal is observed.
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: George Diaz, M.D., Ph.D, Study Director — iECURE, Inc.
Locations (10):
- United States (4):
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - Children's Hospital of Colorado, Anshutz Medical Campus, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Icahn School of Medicine at Mount Sinai, New York, New York
- Australia (2):
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - The Royal Children's Hospital, Melbourne, Victoria
- Spain (2):
  - Hopsital Sant Joan de Deu, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (2):
  - Great Ormond Street Hospital, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust- Great North Children's Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No